CLINICAL TRIAL: NCT02413632
Title: Asymptomatic Sexually Transmitted Infections (STI) : Comparison of Two Screening Strategies Routine Screening Versus Screening as Reported by the Risks Taken by the Patient, in a Cohort of HIV Outpatients Men Who Have Sex With Men
Brief Title: Screening Strategy for Asymptomatic Sexually Transmitted Infections (STI) in a Cohort of HIV Outpatients Men Who Have Sex With Men (DRIVER)
Acronym: DRIVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Collaborators: Saint-Louis Hospital, Paris, France (Other); Bicetre Hospital (Other); Hotel Dieu Hospital (Other); European Georges Pompidou Hospital (Other); Hôpital Necker-Enfants Malades (Other); Hôpital Franco-Britannique (Unknown); Institut Mutualiste Montsouris (Other); Hôpital Lagny Marne la Vallée (Unknown); Hôpital Raymond Poincaré (Other); Centre Hospitalier Argenteuil (Other); Hôpital Louis Mourier (Other); Hospital Ambroise Paré Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 2014/50; 2014-A01358-39 (Other: ANSM)
Record Dates: First submitted 2015-03-07; First posted 2015-04-10 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2017-08

CONDITIONS: HIV
Keywords: HIV-positive MSM (men who have sex with men); asymptomatic sexually transmitted infections; screening
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First period (Other): creation of a STIs score risk
  pharyngeal swab+urinary collection+blood specimens+rectal Chlamydia trachomatis l Neisseria gonorrhoeae (CT/GC) testing
  Interventions: Other: creation of a STIs score risk
- Second period (Other): validation of a STIs score risk
  pharyngeal swab+urinary collection+blood specimens+rectal Chlamydia trachomatis l Neisseria gonorrhoeae (CT/GC) testing
  Interventions: Other: validation of a STIs score risk

INTERVENTIONS:
Other: creation of a STIs score risk — 4 questionnaires 3 screening test ( syphilis, chlamydia, gonorrhea)
  Other Names: First period
  Arms: First period
Other: validation of a STIs score risk — DRIVER questionnaire (DRIVER STI score risk) 3 screening test ( syphilis, chlamydia, gonorrhea)
  Other Names: Second period
  Arms: Second period

SUMMARY:
Comparison of two screening strategies of asymptomatic sexually transmitted infections : routine screening versus screening as reported by the risks taken by the patient, in a cohort of HIV outpatients men who have sex with men. The aim of this study will be create and validate a simple tool for clinicians. A digital tool will be developed will allowed empowerment of HIV-positive men who have sex with men.

DETAILED DESCRIPTION:
Main objectives are :

create and validate a risk score for STIs (DRIVER score) in a population of HIV-positive men who have sex with men (MSM).

determine the prevalence of asymptomatic STIs in a population of HIV-positive MSM

Secondary objectives are :

compare 2 screening strategies regarding STIs in HIV-positive MSM (systematic screening vs screening according to self-declared risk factors) conduct a cost-efficiency analysis of both strategies evaluate patients' knowledge of STIs develop a DRIVER digital tool that will be made available to patients on websites, mobile apps…

Position of the problem :

Over the past 15 years, a resurgence of symptomatic STIs has been observed at both at the global and at the local (French) level. This has been true for gonorrhea since 2008, for syphilis since 2000 and for lymphogranuloma venereum since 2003. The epidemiology of asymptomatic STIs has not been studied as thoroughly but asymptomatic carriage of Neisseria gonorrhoeae and Chlamydia trachomatis as well as latent syphilis account for at least half of cases declared in the past few years. The population of HIV-positive MSM is the demographic category with the highest rates of STIs. In addition, risky sexual attitudes are on the rise in the MSM population in general (in 2010, the French RESIST Network reported that condom use during anal penetrations between males had dropped from 49% in 2008 to 37% in 2010).

Screening practices are currently center- and healthcare-provider dependant. Study will allow a comparison of screening practices thanks to a score that will be built, validated and made available to clinicians and patients.

Type of study : Prospective, non randomized, multicentric and cross-sectional Timeline : Study duration : 18 months Beginning of study : March 2015

ELIGIBILITY:
Inclusion Criteria:

* HIV positive outpatients
* Men who have sex with men
* Speaking, literate french
* Having a french health insurance or an equivalent
* Asymptomatic for a STI the appointment day

Exclusion Criteria:

* Men who never had sex with men
* Protected adults (adults under guardianship)
* Have a STI symptom ( anal discharge, urethritis, proctitis, chancre, rush)

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2015-04; Primary Completion 2017-04-14 (Actual); Study Completion 2017-04-14 (Actual)

PRIMARY OUTCOMES:
Sexually Transmitted Infections risk score in men HIV positive | 6 months
  Construction of a STI risk score

SECONDARY OUTCOMES:
cost-efficacy of a targeted screening versus universal screening | 12 months
  conduct a cost-efficiency analysis of both strategies
patients' knowledge of STIs evaluated by a Sexually Transmitted Disease Knowledge Questionnaire (STD-KQ) | 3 months
  patients' knowledge of STIs will be evaluate
prevalence of asymptomatic STIs in a population of HIV-positive MSM | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David ZUCMAN, MD, Principal Investigator — Hôpital Foch
Locations (17):
- France (17):
  - Hopital Foch, Suresnes, Hauts DE Seine
  - CH Argenteuil, Argenteuil
  - CHU Ambroise Paré, Boulogne-Billancourt
  - CHU Louis Mourier, Colombes
  - Hôpital Raymond Poincaré, Garches
  - CH Marne La Vallée, Jossigny
  - Hôpital Mignot-centre hospitalier de versailles, Le Chesnay
  - CH Bicetre, Le Kremlin-Bicêtre
  - Hôpital Franco-Britannique, Levallois-Perret
  - CHU Necker, Paris
  - Hôtel Dieu, Paris
  - Hôpital de Saint-Antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - CHU St Louis, Paris
  - CHI Poissy/ Saint-Germain en Laye, Saint-Germain-en-Laye
  - CHI Villeneuve Saint-Georges,, Villeneuve-Saint-Georges